CLINICAL TRIAL: NCT00001316
Title: A Study of Viral Burden in Peripheral Blood Versus Lymphoid and Bone Marrow Tissue in People Living With HIV
Brief Title: Viral Load in Blood and Lymph Tissues in People Living With HIV
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 920125; 92-I-0125
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2026-01-20 (Actual); Status verified 2026-01-15

CONDITIONS: HIV
Keywords: Lymph Node; Polymerase Chain Reaction (PCR); In Situ Hybridization; AIDS; Excisional Biopsy; Natural History
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Individuals with HIV: Individuals with HIV
- Individuals without HIV: Individuals without HIV

SUMMARY:
This is a study to determine the effect of the human immunodeficiency virus (HIV) on lymphoid tissues (e.g., lymph nodes) as compared to peripheral white blood cells. We have shown in previous studies that the lymph node is a major site of accumulation of HIV in the body, as well as being a site where much of the viral replication occurs which leads to the destruction of the body's immune system. To better understand the role of the lymph node in HIV infection and destruction of one s immunity, we wish to examine both the virus itself as well as the effects it is having on various types of white cells (called lymphocytes) obtained simultaneously from both peripheral blood and lymph nodes of people living with HIV (PLWH). We also need to look at cells derived from blood and lymph nodes from people who do not have HIV to serve as a control for experiments. We may also use your lymph node tissue and blood cells to attempt to make new T-cells, or rebuild the immune cells, in the laboratory by adding various factors or other substances released by different cells in the body. If you are living with HIV, you may be asked to undergo a second biopsy six weeks to 12 months after the first biopsy. Because of the ability of aspirin to interfere with blood clotting, you must have refrained from the use of aspirin for one week (7 days) prior to the biopsy date. You also cannot use non-aspirin containing, non-steroidal, anti-inflammatory medications (e.g., ibuprofen, naproxen, and similar drugs) one week (7 days) prior to the biopsy. In addition, pregnancy testing will be performed on all females at the time of admission and a positive test will exclude you from participation. No participant will undergo more than six biopsies while participating in this study unless a particular research requires it....

DETAILED DESCRIPTION:
We are studying the pathogenesis of HIV infection and other immune dysfunctions. Because of the lack of an adequate animal model it is generally necessary to utilize human peripheral blood and lymphoid tissues cells for studying aspects of either in vivo or in vitro HIV infection. A dichotomy exists between the amount of HIV that can be measured in peripheral blood compared to lymphoid tissue, as well as the types of immune cells that reside in each compartment. We wish to be able to continue to elucidate many pathogenic aspects of HIV infection and other immune dysfunctions using human peripheral blood mononuclear cells and intact tissue or cells obtained from two major lymphoid organs, lymph nodes and bone marrow.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. HIV status must be documented by a licensed ELISA and confirmed either by Western blot, or plasma viremia.
  2. Aged 18 years or older.
  3. Ability to give informed, written consent.
  4. The following laboratory values:

     1. Absolute neutrophil count of greater than 1000/mm3.
     2. PT, PTT within normal limits (unless PTT is elevated in presence of positive lupus anticoagulant in a participant with no prior history of abnormal bleeding).
     3. Adequate blood counts (PLWH: hemoglobin greater than or equal to 9.0 g/dL, HCT greater than or equal to 28%, platelets greater than or equal to 75,000; participants without HIV: hemoglobin greater than or equal to 11.2 g/dL, HCT greater than or equal to 34.1%, platelets greater than or equal to 150,000).
     4. Blood pressure less than or equal to 180/100; pulse rate 50-100, unless a lower pulse rate is considered normal for the participant.
  5. Participants who do not have HIV will qualify as control participants.
  6. Participants must have a clinically palpable lymph node in an easily accessible location.
  7. Willingness to allow blood samples to be used for future studies of HIV infection/pathogenesis, undergo genetic testing including HLA testing, and undergo hepatitis screening

EXCLUSION CRITERIA:

1. Women who are pregnant and/or breast-feeding.
2. Currently abusing alcohol or other drugs, including narcotics or cocaine.
3. Participants with AIDS dementia or with an AIDS related malignancy other than minimal Kaposi's sarcoma.
4. No Aspirin or Non-Steroidal Anti-inflammatory medications (NSIADs) 7 days prior to procedure. Acetaminophen (Tylenol) is permitted at any time.
5. Any medical condition for which the PI feels LN BX might be contraindicated.
6. Participants in which sedation is planned. Use of narcotics (other than as prescribed by a physician) or cocaine less than 1 week prior to the date of biopsy will be excluded.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Both healthy volunteers and individuals with HIV will be recruited from other existing NIAID studies and from the DC metropolitan area.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 1992-08-26 (Actual)

PRIMARY OUTCOMES:
Relative burden of HIV | Throughout
  The purpose of this project is to determine the relative burden of human immunodeficiency virus (HIV) and/or associated changes in hematopoiesis and immune activation as well as HIV-specific responses in the various subsets of peripheral blood mononuclear cells versus the lymphoid tissues (LT) and bone marrow (BM) in people living with HIV (PLWH).
Immunoregulatory mechanisms | Throughout
  We wish to delineate the precise nature of the immunoregulatory mechanisms and altered homing patterns that contribute to the perturbations in the phenotype and functions of various lymphocyte subsets in peripheral blood versus the lymphoid tissues (LT) of people living with HIV (PLWH).
Effect of Therapy on Viral Burden and Immune Activation | Throughout
  We wish to examine the effect of therapy on viral burden and/or immune activation in the immunoregulatory pathways observed in lymphocyte subsets in lmyphoid tissues (LT) versus peripheral blood mononuclear cells. For LT specimen, the analyses can be performed both on intact tissue sections and excised cells.

CONTACTS AND LOCATIONS:
Overall Officials: Susan L Moir, Ph.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_1992-I-0125.html